CLINICAL TRIAL: NCT01939132
Title: Title of Study: A Single-Site, Investigator Initiated Open-Label Trial of H.P. Acthar Gel (Repository Corticotropin Injection) an Adrenocorticotropic Hormone (ACTH) Analogue in Subjects With Moderately to Severely Active Psoriatic Arthritis (PsA)
Brief Title: Protocol for H.P. Acthar Gel in Moderately to Severely Active Psoriatic Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fiechtner, Justus J., M.D., P.C. (Individual)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02131985
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; ACTH; Acthar
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H.P. Acthar Gel SQ injection (Experimental): Open-label H.P. Acthar Gel 80 units subcutaneously twice weekly for 12 weeks with a 12 week extension.
  Interventions: Drug: Open label H.P. Acthar Gel

INTERVENTIONS:
Drug: Open label H.P. Acthar Gel — Open-label H.P. Acthar Gel 80 units given subcutaneously twice weekly for 12 weeks with 12 week extension.
  Other Names: ACTH

SUMMARY:
Psoriatic arthritis is a heterogeneous chronic inflammatory disorder involving joints, tendon sheaths, entheses, and the axial skeleton as well as skin and nails. This is an open-label trial with H.P. Acthar Gel (80 units/1mL) Subcutaneous injection administered twice weekly. To evaluate the signs and symptoms of psoriatic arthritis after 12 weeks, including American College of Rheumatology 20,Clinical Disease Activity Index, Disease Activity Index 28, Dactylitis and adverse events.

DETAILED DESCRIPTION:
The subjects in this study will be adult men and women ages 18-75 years of age at the time of screening with chronic, moderately-to-severely active PsA and meeting ACR criteria.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, must have adequate reading and writing abilities (in their native language) such that the subject can comprehend and complete the informed consent, and all protocol-related assessments.
2. Age 18-75 years at the time of screening
3. Written informed consent and any locally required authorization (e.g. HIPAA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
4. Subject has had a diagnosis of psoriatic arthritis (by the Classification of Psoriatic Arthritis (CASPAR) criteria) for at least 6 months.
5. Subject must have > 6 tender and >6 swollen joint count at screening.
6. Subject must have > 30 minutes of morning joint stiffness.
7. For subjects receiving non-steroidal anti-inflammatory drugs (NSAIDs) (including PRN use): the subject must be on stable dose for >4 weeks prior to initiation of H.P. Acthar Gel.
8. For subjects receiving any Disease-Modifying Anti-Rheumatic Drug (DMARD) or Biologic agent: subject has received treatment for >8 weeks, with a stable does for > 4 weeks prior to initiation of H.P. Acthar Gel.
9. For subjects receiving oral corticosteroids: the subject must be on a stable dose (not to exceed the equivalent of 10mg of prednisone per day) for >2 weeks prior to initiation of H.P. Acthar Gel.
10. Subject has a negative test for tuberculosis within 6 months before initiating H.P. Acthar Gel defined as either:

    * Negative purified protein derivative (PPD)
    * Negative Quantiferon test, or
    * Negative chest x-ray
11. Females of childbearing potential must use an effective method of birth control and avoid pregnancy from screening through 60 days after final dose of H.P. Acthar Gel unless surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), has a sterile male partner, is >1 year postmenopausal or practices abstinence (not have sexual intercourse):

    -

Exclusion Criteria:

1. Subject has a planned surgical intervention between baseline and the week 24 evaluation.
2. Subject has any concurrent medical condition or uncontrolled, clinically significant systemic disease (eg, renal failure, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency or adrenocortical hyperfunction, peptic ulcer or sensitivity to proteins of porcine origin)
3. Subject has a diagnosis of scleroderma, osteoporosis, fungal infections or ocular herpes simplex
4. History of any type of malignancy <5 years before enrollment into the study (apart from basal cell carcinoma)
5. Any live or attenuated vaccine within 4 weeks prior to signing the informed consent form (administration of killed vaccines is acceptable)
6. Subject has active tuberculosis
7. Any know history of allergy or reaction to any component of H.P. Acthar Gel
8. Known history of a primary immunodeficiency or an underlying condition such as human immunodeficiency virus (HIV) infection.
9. Employees of the clinical study site or any other individuals involved with the conduct of the study or immediate family members of such individuals
10. Concurrent enrollment in any other clinical study with an investigational product within 4 weeks prior to enrollment into the study.
11. Lactating or pregnant females or females who intend to become pregnant anytime from initiation of screening through 60 days post last dose of H.P. Acthar Gel

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
ACR20 (American College of Rheumatology 20) | Week 12
  To evaluate the efficacy of H.P. Acthar Gel given subcutaneously twice weekly on the signs and symptoms of psoriatic arthritis after 12 weeks of administration.
  ACR20 (American College of Rheumatology 20) at week 12

SECONDARY OUTCOMES:
Adverse Events | 24 Weeks
  Adverse events and vital signs will be measured and monitored for 24 weeks.

OTHER OUTCOMES:
Clinical Disease Activity Index (CDAI) | 12 weeks
Disease Activity Index 28 (DAS28) | 12 weeks
Dactylitis (Digit Inflammation) | 12 weeks
  Measure inflammation in fingers and toes

CONTACTS AND LOCATIONS:
Locations (1):
- Justus J. Fiechtner, MD, PC, Lansing, Michigan, United States